CLINICAL TRIAL: NCT06905743
Title: Isometric Contraction-Based Pain Modulation Versus Eccentric Strengthening in Treating Achilles Tendinopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/789
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Contraction-Based Pain Modulation Protocol for Achilles Tendinopathy (Experimental)
  Interventions: Diagnostic Test: Isometric Contraction-Based Pain Modulation Protocol for Achilles Tendinopathy
- Eccentric Strengthening (Alfredson's Protocol for Achilles Tendinopathy ) (Experimental)
  Interventions: Combination Product: Eccentric Strengthening (Alfredson's Protocol for Achilles Tendinopathy )

INTERVENTIONS:
Diagnostic Test: Isometric Contraction-Based Pain Modulation Protocol for Achilles Tendinopathy — The standard recommendation for tendinopathy rehab became 30 to 45 second heavy isometric contractions repeated for 3 to 5 repetitions
  Arms: Isometric Contraction-Based Pain Modulation Protocol for Achilles Tendinopathy
Combination Product: Eccentric Strengthening (Alfredson's Protocol for Achilles Tendinopathy ) — The eccentric loading protocol, popularized by the research of Alfredson, consisted of 3 sets of 15 for both bent knee and straight knee heel raises with each heel lowering lasting 3-seconds
  Arms: Eccentric Strengthening (Alfredson's Protocol for Achilles Tendinopathy )

SUMMARY:
Achilles tendinopathy is a common overuse injury that leads to pain and functional limitations. Traditional rehabilitation focuses on eccentric strengthening, which has been widely studied for its benefits in promoting tendon remodeling and improving strength. However, recent research suggests that isometric contractions may offer superior pain modulation effects, especially in the early stages of rehabilitation.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of isometric contraction-based pain modulation versus eccentric strengthening in treating Achilles tendinopathy. Isometric exercises involve maintaining a static muscle contraction, which has been shown to reduce pain through neuromuscular mechanisms, potentially making it a valuable alternative or complement to eccentric loading.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Diagnosed with Achilles Tendinopathy using MRI
* At least 3 months incidence period of Achilles Tendinopathy
* Must be able to attend all treatment sessions and follow-up assessments.
* Ability to walk independently without any assistive devices.

Exclusion Criteria:

* Severely restricted ROM of ankle
* Patients who underwent surgery for Achilles tendinopathy
* Patients who had undergone previous surgery of lower limb extremity
* Those using ankle orthosis
* Patients with systemic diseases affecting ankle (osteoarthritis, rheumatoid arthritis, and osteoporosis)
* Individuals with neurological disorders affecting the lower limbs.
* Systemic Conditions like diabetes, cardiovascular diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS): | 12 Months
  The Numeric Pain Rating Scale is a widely used, reliable, and user-friendly tool for assessing an individual's level of pain (NPRS). The patient is required to rate their level of discomfort using a self-reported scale with a range of 0 to 10, where ""0"" indicates no pain and ""10"" indicates the most excruciating pain.
PRESSURE ALGOMETRY: | 12 Months
  The pressure pain threshold (PPT), or the lowest force that causes pain in a particular body part, can be objectively measured using pressure algometry. To test sensitivity and identify shifts in pain perception, a portable instrument called a pressure algometer gently and gradually applies pressure to tissue, such as muscles or tendons. Pressure Algometry offers a methodical, objective way to measure pain sensitivity, which is commonly utilized in clinical and research contexts. It is frequently used to evaluate tenderness and pain in musculoskeletal issues, myofascial pain, and tendinopathy. Pressure algometry is a widely used tool to assess mechanical pain sensitivity by applying controlled pressure to a specific area and measuring the pain threshold. Its reliability is well-established, with intra-rater reliability coefficients ranging from 0.70 to 0.94, depending on the site of application and methodological consistency .

CONTACTS AND LOCATIONS:
Locations (1):
- Punjab Social Security Health Management Hospital Manga Raiwind, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No